CLINICAL TRIAL: NCT05584436
Title: The Effect of Follicular Flushing on Oocyte Retrieval Rate and Quality of Embryo Developing From the Index Oocyte: Prospective Cohort Study
Brief Title: The Effect of Follicular Flushing on Oocyte Retrieval Rate and Embryo Quality
Status: Active, not recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, Associate Professor, Akdeniz University
Other Study IDs: 49829697
Record Dates: First submitted 2022-10-06; First posted 2022-10-18 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Infertility
Keywords: oocyte pick up; oocyte retrieval; follicle flushing
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oocytes obtained without flushing: First accessible follicle larger than 12 mm
- oocytes obtained after flushing: Oocytes obtained after a total of 6 cc flushing of follicles that oocyte cumulus complex could not be obtained after the first aspiration

SUMMARY:
Researchers will investigate the effect of flushing according to follicle size on the success of obtaining oocytes from a single follicle. In addition, by comparing the morphological quality of embryos developed from oocytes obtained with and without flushing, the possible effects of flushing on developing embryo quality will be investigated. By evaluating only one follicle for each patient, it is planned to investigate the effectiveness of the flushing process according to individual follicle characteristics, with a study design that has not yet been included in the literature.

DETAILED DESCRIPTION:
Prior to the oocyte pick up (OPU) procedure, the dimensions (height x width x depth) of the first accessible follicle in any ovary will be recorded in millimeters. In this regard, any follicle larger than 12 mm will be selected for the first aspiration. It is planned to evaluate the effectiveness of the washing process in follicles with different sizes by performing the first aspiration procedure regardless of the follicle size. After aspiration of all the follicle fluid with a double lumen needle (17 Gauge), the remaining fluid in the needle and line will be aspirated by giving 2 cc "flushing medium" to the follicle. In this way, all of the pure follicle fluid will be delivered to the in vitro fertilization (IVF) laboratory with the OPU tube for initial evaluation. After the evaluation, if no cumulus oocyte complex (COC) is observed in the first sample, the washing process will be started. In this regard, flushing and aspiration will be performed respectively by giving 2 cc "flushing medium" to the same follicle 3 times. A total of 6 cc flushing medium obtained after the flushing-aspiration process will be delivered to the IVF laboratory and the presence of COC in it will be investigated again under the microscope. Depending on the retrieval of oocyte by direct aspiration or flushing, each oocyte will be followed individually and its quality will be evaluated in case of embryo development from this oocyte.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-43 years old
* Patients who will undergo ICSI procedure

Exclusion Criteria:

* Patients who will undergo oocyte cryopreservation
* Patients with "empty follicle syndrome" in a previous OPU procedure
* Cases that OPU cannot be performed due to premature ovulation

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients between the ages of 18-43 who will undergo OPU between June 2022 and March 2023 will be included in the study.
Sampling Method: Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean number of mature metaphase II oocytes | Through study completion, an average of 1 year
  Number of oocytes that have completed meiosis 1
Mean number of fertilized (2PN) oocytes | Through study completion, an average of 1 year
  Number of oocytes with two pronuclei
Mean number of high-quality blastocyst | Through study completion, an average of 1 year
  Number of embryos with >2BB quality

CONTACTS AND LOCATIONS:
Overall Officials: ŞAFAK OLGAN, MD, Principal Investigator — Akdeniz University; ARİF C ÖZSİPAHİ, MD, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)